CLINICAL TRIAL: NCT03541993
Title: The Cerebral Hemodynamic and Cognitive Effects of Acute Resveratrol Administration in Young, Healthy Adults at 4000 m Stimulated Altitude and at Sea Level: A Double Blind, Crossover Investigation.
Brief Title: The Cerebral Hemodynamic and Cognitive Effects of Acute Resveratrol Administration in Young, Healthy Adults at Stimulated Altitude.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, Tim Eschle, Principal Investigator, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 42AX2
Record Dates: First submitted 2018-04-09; First posted 2018-05-31 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Hypoxia, Altitude; Brain
Keywords: Resveratrol; Cerebral blood flow; Cognition; Hypoxia; Polyphenols
MeSH Terms: conditions — Altitude Sickness; Hypoxia | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Resveratrol Hypoxia (Experimental): 500 mg of trans-resveratrol, tested at a 12.7% atmospheric oxygen level; the equivalent to 4000m above sea level.
  Interventions: Dietary Supplement: Resveratrol
- Placebo Hypoxia (Placebo Comparator): Pharmaceutical grade fumed silica, tested at a 12.7% atmospheric oxygen level; the equivalent to 4000 m above sea level.
  Interventions: Other: Placebo
- Resveratrol Normoxia (Experimental): 500 mg of trans-resveratrol, tested at a 20.9% atmospheric oxygen level; the equivalent to sea level.
  Interventions: Dietary Supplement: Resveratrol
- Placebo Normoxia (Placebo Comparator): Pharmaceutical grade fumed silica, tested at a 20.9% atmospheric oxygen level; the equivalent to sea level.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Resveratrol
  Arms: Resveratrol Hypoxia; Resveratrol Normoxia
Other: Placebo
  Arms: Placebo Hypoxia; Placebo Normoxia

SUMMARY:
Background: Vaso-active polyphenols have been proposed to enhance cognitive performance. Oral administration with the non-flavonoid polyphenol, resveratrol, has been found to modulate cerebral blood flow (CBF); yet, this has not resulted in subsequent predicted benefits to cognitive performance in young, healthy samples. It has been argued that ageing populations who are noted suffer a reduction in CBF and cognition, may possess the subtle deficits to benefit from resveratrol administration. The use of hypoxia has been previously tested by this research group to mimic the decrease in cognitive functioning associated with ageing.

Objectives: The current investigation aimed to further assess if a reduced fraction of inspired oxygen (12.7% FiO2) could provide an experimental model of aging in a young, healthy sample. Moreover, the current study also aimed to assess if resveratrol can attenuate the deficits elicited by the reduction in oxygen supply via increased CBF.

Design: This repeated measures, double blind, placebo controlled, balanced design assessed the cognitive and CBF effects of resveratrol in hypoxia (equivalent to 4000 m above sea level) and normoxia (sea level).

Methods: Twenty-four participants arrived fully fasted (except water) for 12 hours before completing a baseline measure of a cognitive task battery, and taking the treatment for the day (either 500 mg resveratrol or inert placebo). Following a 45 min absorption period, participants completed 3 full repetitions of a cognitive test battery. Changes in cerebral hemodynamics were measured by near-infrared spectroscopy throughout the full testing session.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who provided informed consent.
* Those who didn't meet any of the exclusion criteria.
* Those who took hormonal contraception (e.g.: the pill, coil, implant, etc.) were eligible to participate in the current study.

Exclusion Criteria:

* Individuals below 18 years or above 35 years old at the time of giving consent.
* Individuals with Body Mass Index outside of the range 18-35 kg/m2.
* Individuals with blood pressure greater than 140/90 HH/mg.
* Those who smoke or have smoked.
* Individuals who have been living (for more than 3 months) at an altitude of 2000 m or over within the past 6 months.
* Individuals with a history of neurological, vascular or psychiatric illness (excluding depressive illness and anxiety).
* Individuals with a current diagnosis of depression and/or anxiety.
* Individuals with relevant learning difficulties, dyslexia, dyscalculia or colour blindness.
* Individuals with visual impairment that cannot be corrected with glasses or contact lenses.
* Individuals with frequent migraines that require medication (more than or equal to 1 per month).
* Individuals with disorders of the blood.
* Individuals with a heart disorder.
* Individuals with a respiratory disorder that requires regular medication (Note: asthma sufferers who only take their medication occasionally/as required are eligible for this study).
* Individuals with diabetes.
* Individuals with any food intolerances/sensitivities.
* Females participants who were pregnant, seeking to become pregnant, or currently lactating.
* Individuals currently taking any prescription medications.
* Individuals who have habitually used dietary supplements within the last month (defined as more than 3 consecutive days or 4 days in total).
* Individuals with a history of renal or hepatic disease, or other severe diseases of the gastrointestinal tract (e.g., iron accumulation, iron utilization disorders, hypercalcaemia, hypercalciuria), that are likely to interfere with metabolism/absorption/secretion of the product under investigation.
* Individuals with any health condition that would prevent fulfilment of the study requirements.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-06-07 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2016-12-22 (Actual)

PRIMARY OUTCOMES:
Cerebral blood flow | 2 hours
  Cerebral heamodynamic response (of the prefrontal cortex) was measured at rest and during task performance. The outputs measured here were: oxygenated and deoxygenated haemoglobin concentrations. The addition of these two outputs can also detail total haemoglobin, a proxy for cerebral blood flow. All outputs were reported as concentration change in μmol / L.
Cognitive performance | 1 hour
  Participants completed a number of tasks to measure cognitive performance (as represented by the three main cognitive domains impacted by hypoxia (Memory, Speed of Attention, & Accuracy of Attention)), as part of a 15-minute cognitive battery. Cognitive tasks were scored for accuracy of responses (% correct) and the reaction time to respond to each correct response (in milliseconds (ms)). With the exception of the memory tasks which were scored for the number of correct responses and for the number error responses. Scores across the multiple cognitive tasks were combined to represent the three overall cognitive domains outlined above.